CLINICAL TRIAL: NCT02467257
Title: Potential Role of Gum Arabic as Fetal Hemoglobin Agent in Sudanese Sickle Cell Anemia Patients
Brief Title: Gum Arabic as Fetal Hemoglobin Agent in Sickle Cell Anemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Al-Neelain University (Other)
Collaborators: Military hospital (Unknown); Ministry of Higher Education and Scientific Research, Republic of Sudan (Other Government)
Responsible Party: Principal Investigator, Lamis Kaddam, Dr, Al-Neelain University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AlNeelainU
Record Dates: First submitted 2015-06-04; First posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Gum Arabic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intrevention arm (Experimental): Patients received Gum Arabic as intervention
  Interventions: Dietary Supplement: Gum Arabic

INTERVENTIONS:
Dietary Supplement: Gum Arabic — oral ingestion of 30 gram every day for 12 weeks

SUMMARY:
The purpose of this study is to determine whether Gum Arabic is effective as fetal hemoglobin inducing agent for sickle cell anemia patients.

DETAILED DESCRIPTION:
: High level of fetal haemoglobin (Hb F) decreases sickle cell anaemia (SCA) severity and leads to improved survival. Butyrate proved to increase HbF production in vivo and in vitro studies. Nonetheless, its short half-life limited its utilization in clinical practice. Gum Arabic (GA) is edible, dried, gummy exudate from Acacia Senegal tree. GA fermentation by colonic bacteria increases serum butyrate concentrations. The investigators hypothesized regular intake of GA will increase serum butyrate level. The latter will induce fetal hemoglobin production and ameliorate patients' symptoms. 47 patients hemoglobin SS aged 5-42 years, on regular follow up in Military hospital were recruited from April 2014 to January 2015 Patients received dose of G A 30g/day for 12 weeks. Hb F, complete blood count and Erythropoietin level were measured. The main outcome of interest was the level of HbF after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. over 5 year old
2. less t5han 50
3. diagnosed with homozygous sickle cell anemia by Hb electrophoresis

Exclusion Criteria:

1. patients received blood transfusion within the last three months or admitted to the hospital within 2 weeks because of Sickle cell anemia -related events or crisis.

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study will be the level of fetal hemoglobin after three months | 12 weeks
  fetal hemoglobin will be measured each month for three months

CONTACTS AND LOCATIONS:
Overall Officials: Amal M Saeed, PhD, Study Director — University of Khartoum Faculty of Medicine Department of Physiology; Lamis AA Kaddam, MSc, Principal Investigator — Department of physiology Faculty of Medicine Alneelain University Khartoum,
Locations (1):
- Military Hospital, Omdurman, Khartoum State, Sudan

REFERENCES:
- [Background] Fathallah H, Atweh GF. Induction of fetal hemoglobin in the treatment of sickle cell disease. Hematology Am Soc Hematol Educ Program. 2006:58-62. doi: 10.1182/asheducation-2006.1.58. PMID 17124041
- [Background] Kutlar A, Reid ME, Inati A, Taher AT, Abboud MR, El-Beshlawy A, Buchanan GR, Smith H, Ataga KI, Perrine SP, Ghalie RG. A dose-escalation phase IIa study of 2,2-dimethylbutyrate (HQK-1001), an oral fetal globin inducer, in sickle cell disease. Am J Hematol. 2013 Nov;88(11):E255-60. doi: 10.1002/ajh.23533. Epub 2013 Oct 3. PMID 23828223
- [Background] Matsumoto N, Riley S, Fraser D, Al-Assaf S, Ishimura E, Wolever T, Phillips GO, Phillips AO. Butyrate modulates TGF-beta1 generation and function: potential renal benefit for Acacia(sen) SUPERGUM (gum arabic)? Kidney Int. 2006 Jan;69(2):257-65. doi: 10.1038/sj.ki.5000028. PMID 16408114
- [Background] Ballal A, Bobbala D, Qadri SM, Foller M, Kempe D, Nasir O, Saeed A, Lang F. Anti-malarial effect of gum arabic. Malar J. 2011 May 20;10:139. doi: 10.1186/1475-2875-10-139. PMID 21599958
- [Derived] Kaddam LA, Kaddam AS. Effect of Gum Arabic (Acacia senegal) on C-reactive protein level among sickle cell anemia patients. BMC Res Notes. 2020 Mar 18;13(1):162. doi: 10.1186/s13104-020-05016-2. PMID 32188508
- [Derived] Kaddam L, Fadl-Elmula I, Eisawi OA, Abdelrazig HA, Saeed AM. Acacia Senegal (Gum Arabic) Supplementation Modulate Lipid Profile and Ameliorated Dyslipidemia among Sickle Cell Anemia Patients. J Lipids. 2019 Jun 18;2019:3129461. doi: 10.1155/2019/3129461. eCollection 2019. PMID 31316836
- [Derived] Kaddam LA, Fdl-Elmula I, Eisawi OA, Abdelrazig HA, Elnimeiri MK, Saeed AM. Biochemical effects and safety of Gum arabic (Acacia Senegal) supplementation in patients with sickle cell anemia. Blood Res. 2019 Mar;54(1):31-37. doi: 10.5045/br.2019.54.1.31. Epub 2019 Mar 21. PMID 30956961
- [Derived] Kaddam L, Fadl-Elmula I, Eisawi OA, Abdelrazig HA, Salih MA, Lang F, Saeed AM. Gum Arabic as novel anti-oxidant agent in sickle cell anemia, phase II trial. BMC Hematol. 2017 Mar 16;17:4. doi: 10.1186/s12878-017-0075-y. eCollection 2017. PMID 28331623
- [Derived] Kaddam L, FdleAlmula I, Eisawi OA, Abdelrazig HA, Elnimeiri M, Lang F, Saeed AM. Gum Arabic as fetal hemoglobin inducing agent in sickle cell anemia; in vivo study. BMC Hematol. 2015 Dec 29;15:19. doi: 10.1186/s12878-015-0040-6. eCollection 2015. PMID 26719803